CLINICAL TRIAL: NCT04370314
Title: Clinical Performance of One-piece Screw-retained Implant Crowns Base on CAD/CAM Hand-veneered Zirconium Dioxide Customized Abutments With a 6 Years and 7 Months Mean Follow-up
Brief Title: Retrospective Study on Clinical Performance of Screw-retained Implant Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020/13
Record Dates: First submitted 2020-04-24; First posted 2020-04-30 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Dental Implant Failed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zirconia implant-supported crown (Experimental): Full zirconia implant-supported crown
  Interventions: Other: Dental prosthetics

INTERVENTIONS:
Other: Dental prosthetics — Implant-supported crowns

SUMMARY:
Survival and success rates of all-ceramic implant-supported fixed reconstructions fabricated with CAD/CAM technology after at least one year in function.

Survival and success rates (clinical, radiologic and esthetic) of all-ceramic implant-supported fixed reconstructions fabricated with CAD/CAM technology after 2 to 10 years in function.

Establishment of a database of patients with all-ceramic implant-supported fixed reconstructions fabricated with CAD/CAM technology for future longitudinal retrospective studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one fixed all-ceramic reconstruction (single implant restoration on BL implant with individualized zirconia abutment directly screwed and directly veneered, three- to five-unit zirconia bridges directly veneered, single tooth crown made of a lithium disilicate glass-ceramic (LS2) blank)
* Written informed consent

Exclusion Criteria:

* Pregnancy at the time of the follow-up examination
* Mental handicap
* Patients that could not be contacted/located
* Patients not interested in participating
* Patients with the need of antibiotic prophylaxis prior to a clinical examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Survival and success rates of all-ceramic implant-supported fixed reconstructions | 1 year
  Number of all-ceramic implant-supported fixed reconstructions fabricated with CAD/CAM technology still in place after at least one year in function.

SECONDARY OUTCOMES:
Number of patients with biological complications assessed via clinical examination | 1 year
  A clinical evaluation of the implant crowns will be performed in order to detect any kind of biological complication, namely periimplantitis and perimucositis
Number of patients with biological complications assessed via periapical x-ray | 1 year
  A radiological evaluation of the implant crowns will be performed to measure and evaluate the bone crestal changes
Number of patients with technical complications | 1 year
  A clinical evaluation of the implant crowns will be performed in order to detect any kind of complication, namely chipping, screw loosening or abutment fracture
Patient satisfaction as assessed by VAS A | 1 year
  Patients assess by patient questionnaire their implant reconstructions, in terms of function by means of a Visual Analog Scale (VAS A), where the parameter will be scored from 1 to 10.
Patient satisfaction as assessed by VAS B | 1 year
  Patients assess by patient questionnaire their implant reconstructions, in terms of esthetics by means of a Visual Analog Scale (VAS B), where the parameter will be scored from 1 to 10.
Esthetic outcome | 1 year
  The esthetic examination included the Pink and White Esthetic Score Assessment (PES/WES) according to Belser et al. 2009 & Furhäuser et al. 2005 on a scale from 0-10 whereas 10 means an optimal outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Manrique Fonseca, Dr., Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fonseca M, Molinero-Mourelle P, Forrer FA, Schnider N, Hicklin SP, Schimmel M, Bragger U. Clinical performance of implant crowns with customized zirconia abutments: A prospective cohort study with a 4.5- to 8.8-year follow-up. Clin Oral Implants Res. 2021 Jul;32(7):853-862. doi: 10.1111/clr.13761. Epub 2021 May 24. PMID 33949004